CLINICAL TRIAL: NCT01397487
Title: Effects of the Blastomere Biopsy of Day 3 Human Embryos on Blastocyst Percentage, Cell Number of Obtained Blastocyst and Implantation Rate
Brief Title: Effects of Day 3 Blastomere Biopsy on Human Embryos
Acronym: BB
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Para La Investigacion Hospital La Fe (Other)
Responsible Party: FUNDACION PARA LA INVESTIGACION HOSPITAL LA FE, Hospital Universitari y Politecnic La Fe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/0416
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Blastomere Biopsy Safety
Keywords: morphometric parameters, embryo biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one single arm (Other): All patients are included to complete a biopsy of half part of the embryos
  Interventions: Procedure: Blastomere biopsy

INTERVENTIONS:
Procedure: Blastomere biopsy — The blastomere biopsy will be done after 72 hours of embryo culture. An inverted microscope Olympus IX70 with a heated stage will be used to perform the biopsy. The micromanipulation for the blastomere extraction will be made with a micropipette MBB-FP-M-30 (Humagen).

SUMMARY:
The aim of this study to evaluate the effect of embryo biopsy on blastocyst development and implantation rate.

DETAILED DESCRIPTION:
Preimplantation genetic diagnosis (PGD) was initially developed to prevent monogenic diseases. However, its use has been extended to improve pregnancy rates in assisted reproductive techniques (ART). These new indications has been called screening for aneuploidy (PGS, preimplantation genetic screening). The current indications for PGS include advanced maternal age, recurrent miscarriage, repeated implantation failure, severe male factor infertility, previous aneuploid pregnancy, poor embryo quality, chemotherapy and radiotherapy and elective single embryo transfer to avoid multiple pregnancies. Nevertheless, the results obtained in the last decade have failed to clearly demonstrate any benefit of PGS in these indications and there are no studies evaluating the effect that biopsy could produce on embryos.

Markers of embryo quality are still very limited and are based on subjective morphological parameters (such as cell number, size and degree of fragmentation) or on the study of embryonic development by measuring the percentage of embryos reaching the blastocyst stage after 120 hours of in vitro culture. Counting the cell number of blastocysts involves the staining and subsequent nuclei counting, which is incompatible with later embryo transfer. A valid alternative to avoid nuclear staining would be a morphometric study using optical sections of different focal planes of the blastocyst and three dimensional (3D) virtual reconstructions.

ELIGIBILITY:
Inclusion Criteria:

* No relevant medical history.
* BMI < 25.
* Age < 35 years old.
* Unexplained infertility, tubal or male cause of infertility.
* Between 6 and 8 embryos on day 3 of embryo culture.

Exclusion Criteria:

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-01 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Blastocyst percentage | after 120 hours of culture

SECONDARY OUTCOMES:
Number of cells of blastocyst measured by morphometric analysis | after 120 hours of culture
Implantation rate | after one month of embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pellicer, MDPhD, Study Director — La Fe Hospital. Dept. of Obstetrics and Gynecology.; Amparo Mercader, P.h.D, Study Chair — Instituto Valenciano de Infertilidad. PGD Laboratory.
Locations (1):
- La Fe University Hospital. Department of Obstetrics and Gynecology, Valencia, Valencia, Spain